CLINICAL TRIAL: NCT03216863
Title: Home Respiratory Rehabilitation in Patients With Lung Cancer Non-small Cell Advanced or Metastatic Treated With Oral Targeted Therapy
Brief Title: Home Respiratory Rehabilitation in Advanced Lung Cancer Chemotherapy Per os
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014_61; 2015-A00468-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with advanced or metastatic non-small cell lung cancer treated with oral targeted therapy (tyrosine kinase (TKI) inhibitors of EGF-R and ALK inhibitors), regardless of the treatment line.
Oversight: Data Monitoring Committee: No

ARMS (1):
- 8 weeks Respiratory rehabilitation (Experimental)
  Interventions: Other: Respiratory rehabilitation

INTERVENTIONS:
Other: Respiratory rehabilitation — It consists of a global care of the patient: therapeutic education, nutritional maintenance, psychological support and re-training to the effort at home after discharge or after follow up visit of targeted therapy

SUMMARY:
The feasibility and impact of respiratory rehabilitation (RR) in patients with advanced or metastatic (EGF-R WT or mutated) non-small cell lung cancer treated with oral targeted therapy including Inhibitors of EGF-R tyrosine kinases (TKI) and ALK inhibitors.

These patients will benefit, at the beginning of the chemotherapy whatever the treatment line, of a respiratory rehabilitation. The respiratory rehabilitation takes place at the patient's home with the HAD's cooperation 3 hours per week, divided into 2 or 3 sessions. There is associated educational, nutritional and psychological support for a total duration of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient with advanced or metastatic lung cancer
* In the course of treatment by oral chemotherapy of oral targeted therapy (tyrosine kinase inhibitor) in 1st, 2nd, 3rd line or more at the time of their inclusion
* Diagnosis of CP retained after multidisciplinary discussion of patient records

Exclusion Criteria:

* Any residual toxicity of a previous antineoplastic treatment, grade> 2.
* Cardio-respiratory contraindications to exercise re-training:
* Angina unstable
* Recent infarct
* Tight aortic stenosis
* Unsteady heart failure
* Pericarditis, endocarditis, myocarditis
* Evolutionary thromboembolic disease
* Ventricular aneurysm
* Intra ventricular thrombus
* Uncontrolled rhythm disorders
* Instability of the respiratory state defined by uncompensated respiratory acidosis
* Carcinological contraindications:
* Bone metastases at risk of fracture and / or algae despite optimal analgesic treatment, symptomatic central nervous system metastases
* Presence of anemia (Hb <8g / dl or <10g / dl if patient with previous cardiac history), thrombocytopenia (<100,000 platelets / mm3)
* Chimio toxicity (neurological, cardiac) according to the investigator's assessment
* Neuromuscular contraindications:
* Neuromuscular and / or osteo-articular disease making it impossible to re-train
* Severe cognitive impairment
* Patient under tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Rate of patients completing the full Respiratory Rehabilitation (8 weeks) at home | At 8 weeks

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy Lung standardized | Baseline and 8 weeks
  measure the quality of life
EORTC QLQ C-30 standardized version 3.0 | Baseline and 8 weeks
  Measure the quality of life
Functional capacity | Baseline and 8 weeks
  Exercise capacity with the six minutes walk test
Respiratory capacity | Baseline and 8 weeks
  measured by the spirometry
Nutritional Risk Screening score | Baseline and 8 weeks
  Nutritional state assessment by albumine and pre albumine dosage
Body Mass Index | Baseline and 8 weeks
Overall and progression-free survival | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Scherpereel, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (3):
- France (3):
  - Hôpital Calmette, CHRU, Lille
  - Hôpital privé La Louvière, Lille
  - Centre hospitalier Victor Provo, Roubaix

IPD SHARING:
Plan to Share IPD: No